CLINICAL TRIAL: NCT02099058
Title: A Multicenter, Phase 1/1b, Open-Label, Dose-Escalation Study of ABBV-399, an Antibody Drug Conjugate, in Subjects With Advanced Solid Tumors
Brief Title: A Study Evaluating the Safety, Pharmacokinetics (PK), and Preliminary Efficacy of ABBV-399 in Participants With Advanced Solid Tumors
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: M14-237; 2014-003154-14 (EudraCT Number)
Record Dates: First submitted 2014-03-26; First posted 2014-03-28 (Estimated); Last update posted 2025-08-14 (Actual); Status verified 2025-08

CONDITIONS: Advanced Solid Tumors Cancer
Keywords: Cancer; Advanced Solid Tumor; Neoplasm
MeSH Terms: conditions — Neoplasms | interventions — osimertinib; Nivolumab; telisotuzumab vedotin; Erlotinib Hydrochloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (6):
- Monotherapy Telisotuzumab vedotin (21-day dosing cycles) (Experimental): Telisotuzumab vedotin will be administered at escalating dose levels in 21-day dosing cycles. Additional subjects will be enrolled in an expansion cohort that will further evaluate Telisotuzumab vedotin.
  Interventions: Drug: Telisotuzumab vedotin
- Monotherapy Telisotuzumab vedotin(28-day dosing cycles) (Experimental): Telisotuzumab vedotin will be administered at escalating dose levels in 28-day dosing cycles. Additional subjects will be enrolled in an expansion cohort that will further evaluate Telisotuzumab vedotin.
  Interventions: Drug: Telisotuzumab vedotin
- Monotherapy Expansion Cohort (Experimental): Telisotuzumab vedotin will be administered every 14 days on a 28-day dosing cycle.
  Interventions: Drug: Telisotuzumab vedotin
- Arm A (Telisotuzumab vedotin plus Erlotinib) (Experimental): Telisotuzumab vedotin to be evaluated with Erlotinib.
  Interventions: Drug: Telisotuzumab vedotin; Drug: Erlotinib
- Arm D (Telisotuzumab vedotin plus Nivolumab) (Experimental): Telisotuzumab vedotin to be evaluated with Nivolumab.
  Interventions: Drug: Nivolumab; Drug: Telisotuzumab vedotin
- Arm E (Telisotuzumab vedotin plus Osimertinib) (Experimental): Telisotuzumab vedotin to be evaluated with Osimertinib.
  Interventions: Drug: Osimertinib; Drug: Telisotuzumab vedotin

INTERVENTIONS:
Drug: Osimertinib — It is administered orally everyday.
  Arms: Arm E (Telisotuzumab vedotin plus Osimertinib)
Drug: Nivolumab — It is an intravenous infusion administered every 14 days.
  Arms: Arm D (Telisotuzumab vedotin plus Nivolumab)
Drug: Telisotuzumab vedotin — It is administered by infusion in 21-day dosing cycles.
  Other Names: ABBV-399
  Arms: Arm A (Telisotuzumab vedotin plus Erlotinib); Monotherapy Telisotuzumab vedotin (21-day dosing cycles)
Drug: Telisotuzumab vedotin — It is administered by infusion in 28-day dosing cycles.
  Other Names: ABBV-399
  Arms: Arm D (Telisotuzumab vedotin plus Nivolumab); Arm E (Telisotuzumab vedotin plus Osimertinib); Monotherapy Expansion Cohort; Monotherapy Telisotuzumab vedotin(28-day dosing cycles)
Drug: Erlotinib — It is administered orally everyday.
  Arms: Arm A (Telisotuzumab vedotin plus Erlotinib)

SUMMARY:
This is a Phase 1/1b open-label study evaluating the safety, pharmacokinetics (PK), and preliminary efficacy of ABBV-399 as monotherapy and in combination with osimertinib, erlotinib, and nivolumab in participants with advanced solid tumors likely to express c-Met. Enrollment is closed for the monotherapy arms, Arm A, and Arm D.

ELIGIBILITY:
Inclusion Criteria:

* Participant must have advanced Non-Small Cell Lung Cancer (NSCLC) that is not amenable to surgical resection or other approved therapeutic options that have demonstrated clinical benefit.
* Participant has an Eastern Cooperative Oncology Group (ECOG) Performance Status of 0 to 2. For Monotherapy Expansion Cohort, participant must have ECOG Performance Status of 0 or 1.
* Participant must have measurable disease per Response Evaluation Criteria In Solid Tumors (RECIST) version 1.1.
* Participant has archived diagnostic formalin-fixed paraffin embedded (FFPE) tumor tissue confirmed available for analyses.
* Participant has adequate bone marrow, renal, and hepatic function.
* Women of childbearing potential must have a negative serum pregnancy test at baseline.
* Participants in the combination therapy arms A and D must be eligible to receive erlotinib, or nivolumab per most locally approved labeling, or at the discretion of the Investigator.
* Participants in the combination therapy Arm E must satisfy following criteria.

  * Participant must have metastatic/locally advanced nonsquamous NSCLC with documented Epidermal Growth Factor Receptor (EGFR) mutation(s) del19 or L858R, with or without T790M mutation, and none of the EGFR mutations known to be resistant to osimertinib.
  * Participant must have received at least 1 but no more than 2 prior regimens, one of which must have contained osimertinib. Participant must have had disease progression while on osimertinib. Only 1 prior regimen may have contained chemotherapy. Consecutive EGFR TKIs will count as 1 regimen
  * Participant must have available post-progression tumor tissue for central c-Met immunohistochemistry (IHC) testing.
  * Participant has adequate bone marrow function.
* Participants in the Monotherapy Expansion Cohort must satisfy following criteria.

  * Participant must have locally advanced or metastatic, non-squamous, EGFR wild type, c-Met+ NSCLC. Participants must not have adenosquamous histology.
  * Participant must have received no more than 2 lines of prior systemic therapy (including no more than 1 line of systemic cytotoxic chemotherapy) in the locally advanced or metastatic setting.
  * Participant must have progressed on systemic cytotoxic chemotherapy (or are ineligible for systemic cytotoxic chemotherapy) and an immune checkpoint inhibitor (as monotherapy or in combination with systemic cytotoxic chemotherapy, or ineligible for an immune checkpoint inhibitor), and prior anti-cancer therapies targeting driver gene alterations (if applicable).
  * Participant should not have received prior c-Met-targeted antibody-based therapies.

Exclusion Criteria:

* Participant has received radiation therapy to the lung < 6 months prior to the first dose of ABBV-399.
* Participant has received anticancer therapy including chemotherapy, immunotherapy, biologic, or any investigational therapy within a period of 21 days or herbal therapy within 7 days prior to the first dose of ABBV-399.
* Participant has uncontrolled metastases to the central nervous system (CNS) based on head CT or MRI. Participants with brain metastases may be eligible 2-4 weeks after definitive therapy to all known sites of CNS disease provided they are asymptomatic and either off or on a non-increasing dose (in last 2 weeks) of systemic steroids and not on anticonvulsants for seizure activity directly related to progressive CNS metastases.
* Participant has history of interstitial lung disease (ILD) or pneumonitis that required treatment with systemic steroids.
* Participant has evidence of pulmonary fibrosis on screening imaging assessment or any history of pneumonitis or interstitial lung disease (ILD) within 3 months of the planned first dose of the study drug.
* Participant has unresolved clinically significant adverse events >= Grade 2 from prior anticancer therapy, except for alopecia or anemia.
* Participant has had major surgery within 21 days prior to the first dose of ABBV-399.
* Participant has a clinically significant condition(s) described in the protocol.
* History of major immunologic reaction to any Immunoglobulin G (IgG) containing agent.
* Participant has any medical condition which in the opinion of the Investigator or Medical Monitor places the participant at an unacceptably high risk for toxicities.
* Participant is a lactating or pregnant female.
* Participant with known active COVID-19 infection, subjects with signs/symptoms associated with COVID-19 infection or known exposure to a confirmed case of COVID-19 infection during 14 days prior to Screening must be screen failed and may only rescreen after they have recovered from COVID-19 and they are no longer considered contagious, per investigator assessment.
* Participants enrolled on the combination therapy phase must satisfy the above exclusion criteria and also the following:

  * Participants may not receive ABBV-399 in combination with osimertinib, erlotinib or nivolumab if they have any medical condition which in the opinion of the Investigator places the participant at an unacceptably high risk for toxicities from the combination.
  * Participants may not receive nivolumab if they have:

    * Active autoimmune disease with exceptions of vitiligo, type I diabetes mellitus, hypothyroidism and psoriasis.
    * Used systemic corticosteroids (> 10 mg daily prednisone or equivalent) or other immunosuppressive medications within 14 days of study drug administration, with exception of inhaled, locally injected or topical steroids.
    * Known immunosuppressive disease, for example human immunodeficiency virus infection or history of bone marrow transplant or chronic lymphocytic leukemia.
  * Participants may not be enrolled into the osimertinib Combination Therapy Arm E if they have the following:

    * History of hypersensitivity to active or inactive excipients of osimertinib.
    * History of osimertinib dose reduction.
    * Refractory nausea and vomiting, chronic gastrointestinal diseases, inability to swallow the formulated product, or previous significant bowel resection that would preclude adequate absorption of osimertinib.
    * Any of the following cardiac criteria: a) Mean resting corrected QT interval (QTc) > 470 ms; b) Any clinically important abnormalities in rhythm, conduction, or morphology of resting ECG, e.g., complete left bundle branch block, second- or third-degree heart block, PR interval > 250 ms; c) Any factors that increase the risk of QTc prolongation or risk of arrhythmic events such as heart failure, hypokalemia, congenital long QT syndrome, or any concomitant medication known to prolong the QT interval.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 237 (Actual)
Dates: Start 2014-01-15 (Actual); Primary Completion 2026-08 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
Number of Participants with Adverse Events | Up to 24 Months
  An adverse event (AE) is defined as any untoward medical occurrence in a patient or clinical investigation subject administered a pharmaceutical product and which does not necessarily have a causal relationship with this treatment.
Recommended Phase 2 Dose (RPTD) of ABBV-399 when Administered as Monotherapy and in Combination with Osimertinib, Erlotinib or Nivolumab | Up to 24 Months
  The RPTD of ABBV-399 when administered as monotherapy and in combination with osimertinib, erlotinib or nivolumab will be determined during the dose escalation phase of the study. RPTD will be determined using available safety and pharmacokinetics data.
Area under the curve (AUC) from time zero to the last measurable concentration AUC (0-t) | Up to 24 months
  AUC (0-t) = Area under the serum concentration versus time curve from time zero (pre-dose) to the time of the last measurable concentration.
Maximum observed plasma concentration (Cmax) | Up to 24 months
  Maximum observed plasma concentration (Cmax).
Time to Cmax (Tmax) | Up to 24 months
  Time to Cmax (Tmax).
Terminal elimination half life | Up to 24 months
  Terminal elimination half life.

CONTACTS AND LOCATIONS:
Overall Officials: ABBVIE INC., Study Director — AbbVie
Locations (36):
- United States (21):
  - Scottsdale Healthcare /ID# 123761, Scottsdale, Arizona
  - City of Hope /ID# 153759, Duarte, California
  - University of California, Los Angeles /ID# 148295, Los Angeles, California
  - UC Irvine /ID# 165107, Orange, California
  - University of California, Davis Comprehensive Cancer Center /ID# 129805, Sacramento, California
  - Univ of Colorado Cancer Center /ID# 123759, Aurora, Colorado
  - The University of Chicago Medical Center /ID# 136995, Chicago, Illinois
  - Ingalls Memorial Hosp /ID# 165876, Harvey, Illinois
  - Massachusetts General Hospital /ID# 129804, Boston, Massachusetts
  - Dana-Farber Cancer Institute /ID# 168782, Boston, Massachusetts
  - Duplicate_Henry Ford Health System /ID# 149857, Detroit, Michigan
  - Herbert Herman Cancer Center /ID# 149858, Lansing, Michigan
  - Washington University-School of Medicine /ID# 143798, St Louis, Missouri
  - Summit Medical Group-Florham Park /ID# 217651, Florham Park, New Jersey
  - Northwell Health - Monter Cancer Center /ID# 218170, Lake Success, New York
  - Montefiore Medical Park at Eastchester /ID# 218445, The Bronx, New York
  - Duke Cancer Center /ID# 123763, Durham, North Carolina
  - Tennessee Oncology, PLLC /ID# 129802, Nashville, Tennessee
  - Mary Crowley Cancer Research /ID# 123760, Dallas, Texas
  - University of Texas MD Anderson Cancer Center /ID# 154648, Houston, Texas
  - Virginia Cancer Specialists - Fairfax /ID# 165708, Fairfax, Virginia
- Universitair Ziekenhuis Antwerpen /ID# 170118, Edegem, Antwerpen, Belgium
- Duplicate_Tampere University Hospital /ID# 165065, Tampere, Pirkanmaa, Finland
- France (2):
  - AP-HM - Hopital de la Timone /ID# 151570, Marseille, Bouches-du-Rhone
  - Institut Gustave Roussy /ID# 132747, Villejuif, Val-de-Marne
- Duplicate_Istituto Romagnolo per lo Studio dei Tumori "Dino Amadori" - IRCCS /ID# 164077, Meldola, Emilia-Romagna, Italy
- Japan (2):
  - National Cancer Center Hospital East /ID# 217570, Kashiwa-shi, Chiba
  - National Cancer Center Hospital /ID# 217571, Chuo-ku, Tokyo
- Radboud Universitair Medisch Centrum /ID# 246908, Nijmegen, Gelderland, Netherlands
- South Korea (3):
  - Duplicate_The Catholic University of Korea, ST. Vincent's Hospital /ID# 233378, Suwon, Gyeonggido
  - Asan Medical Center /ID# 217334, Seoul, Seoul Teugbyeolsi
  - Yonsei University Health System Severance Hospital /ID# 217333, Seoul
- Taiwan (4):
  - China Medical University Hospital /ID# 217494, Taichung, Taichung
  - National Cheng Kung University Hospital /ID# 167175, Tainan, Tainan
  - National Taiwan University Hospital /ID# 167173, Taipei City, Taipei
  - Taipei Veterans General Hosp /ID# 217392, Taipei, Taipei

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Camidge DR, Barlesi F, Goldman JW, Morgensztern D, Heist R, Vokes E, Spira A, Angevin E, Su WC, Hong DS, Strickler JH, Motwani M, Dunbar M, Parikh A, Noon E, Blot V, Wu J, Kelly K. Phase Ib Study of Telisotuzumab Vedotin in Combination With Erlotinib in Patients With c-Met Protein-Expressing Non-Small-Cell Lung Cancer. J Clin Oncol. 2023 Feb 10;41(5):1105-1115. doi: 10.1200/JCO.22.00739. Epub 2022 Oct 26. PMID 36288547
- [Derived] Camidge DR, Morgensztern D, Heist RS, Barve M, Vokes E, Goldman JW, Hong DS, Bauer TM, Strickler JH, Angevin E, Motwani M, Parikh A, Sun Z, Bach BA, Wu J, Komarnitsky PB, Kelly K. Phase I Study of 2- or 3-Week Dosing of Telisotuzumab Vedotin, an Antibody-Drug Conjugate Targeting c-Met, Monotherapy in Patients with Advanced Non-Small Cell Lung Carcinoma. Clin Cancer Res. 2021 Nov 1;27(21):5781-5792. doi: 10.1158/1078-0432.CCR-21-0765. Epub 2021 Aug 23. PMID 34426443
- [Derived] Strickler JH, Weekes CD, Nemunaitis J, Ramanathan RK, Heist RS, Morgensztern D, Angevin E, Bauer TM, Yue H, Motwani M, Parikh A, Reilly EB, Afar D, Naumovski L, Kelly K. First-in-Human Phase I, Dose-Escalation and -Expansion Study of Telisotuzumab Vedotin, an Antibody-Drug Conjugate Targeting c-Met, in Patients With Advanced Solid Tumors. J Clin Oncol. 2018 Nov 20;36(33):3298-3306. doi: 10.1200/JCO.2018.78.7697. Epub 2018 Oct 4. PMID 30285518